CLINICAL TRIAL: NCT01576666
Title: A Phase Ib, Multi-center, Open Label, Dose Escalation Study of Oral LDE225 in Combination With BKM 120 in Patients With Advanced Solid Tumors
Brief Title: Phase Ib, Dose Escalation Study of Oral LDE225 in Combination With BKM120 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CLDE225X2114; 2011-005016-28 (EudraCT Number)
Record Dates: First submitted 2012-04-10; First posted 2012-04-12 (Estimated); Last update posted 2020-12-19 (Actual); Status verified 2016-02

CONDITIONS: Dose Escalation; Safety; Preliminary Efficacy; Advanced Solid Tumors; Metastatic Breast Cancer; Advanced Pancreatic Adenocarcinoma; Metastatic Colorectal Cancer; Recurrent Glioblastoma Multiforme; Gastric Cancer; Gastroesophageal Junction Cancer; Triple Negative Metastatic Breast Cancer; Hormone Receptor Positive (ER+/PR+, and Her2-) Metastatic Breast Cancer
Keywords: Dose escalation; Maximum Tolerated Dose; MTD; Safety Expansion; Safety; Preliminary Efficacy; Objective Response Rate; Early progression rate; PI3K activation; Combination Treatment; Hedgehog Signaling Pathway; Smoothened inhibitor; Phosphoinositide-3' kinase; Phosphatase signaling pathway; Advanced solid tumors; metastatic breast cancer; advanced pancreatic adenocarcinoma; metastatic colorectal cancer; recurrent glioblastoma multiforme; gastric cancer; gastroesophageal junction cancer; triple negative metastatic breast cancer; hormone receptor positive (ER+/PR+, and Her2-) metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Glioblastoma; Stomach Neoplasms | interventions — sonidegib; NVP-BKM120

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LDE225 and BKM120 in combination (Experimental): LDE225 and BKM120 in combination
  Interventions: Drug: LDE225; Drug: BKM120

INTERVENTIONS:
Drug: LDE225
Drug: BKM120

SUMMARY:
The purpose of this study is to determine the maximum dose of LDE225 and BKM120 that can be safely given together to patients and/or the dose that will be used in future studies. This study will also learn more about how the combination of these two investigational drugs may work for patients with certain cancers (specifically metastatic breast cancer, advanced pancreatic adenocarcinoma, metastatic colorectal cancer and recurrent glioblastoma multiforme).

DETAILED DESCRIPTION:
The primary purpose of this study is to determine a combination maximum tolerated dose (MTD) and/or recommended dose for expansion (RDE) of LDE225 and BKM120 when co-administered orally in patients with advanced solid tumors. Adult patients, aged > 18 years with advanced solid tumors that have progressed despite standard therapy or for which no standard therapies exist will be eligible for this study.

In the dose escalation part of the study, four groups of patients with the following tumor types will be enrolled: recurrent GBM, metastatic breast cancer, metastatic CRC and advanced pancreatic adenocarcinoma. It is anticipated that approximately 45 patients will be enrolled in the dose escalation part. Approximately 15 GBM patients (maximum of 2 patients per dose level) will be enrolled to previously well-tolerated doses during dose escalation if no slot is available in a cohort under active testing. In the dose expansion part of the study, five groups of patients (approximately 15 patients per group) with the following tumor types will be enrolled: recurrent GBM, triple negative metastatic breast cancer, hormone receptor positive (ER+/PR+, and Her2-) metastatic breast cancer, gastric/gastroesophageal junction cancer, and a combined maximum of 15 patients with metastatic CRC or advanced pancreatic adenocarcinoma. The dose expansion will enroll approximately 75 patients. Accounting for patients who may withdraw or who may not meet the eligibility criteria, it is expected that this study will enroll approximately 120 patients.

This is a multi-center, open-label, dose finding, phase Ib study to determine the MTD and/or RDE for the combination of LDE225 plus BKM120, followed by an expansion part to further assess safety and preliminary efficacy of the combination in patients with advanced solid tumors that are frequently associated with dysregulated Hh and/or PI3K pathways, specifically triple negative metastatic breast cancer, hormone receptor positive (ER+/PR+, and Her2-) metastatic breast cancer, advanced pancreatic adenocarcinoma, metastatic CRC, recurrent GBM and gastric/gastroesophageal junction cancer patients. Patients will be treated daily on 28-day cycles. Dose escalation will be dependent on the available toxicity information (including adverse events that are not DLTs), PK, PD, and efficacy information, as well as the recommendations from the Bayesian Logistic Regression Model (BLRM).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adult patients (> 18 years)
2. Patients with histologically/cytologically confirmed diagnosis of the following advanced tumors that have progressed despite standard therapy or that have no available established treatments: metastatic breast cancer, pancreatic adenocarcinoma, metastatic CRC or recurrent GBM will be included.
3. Provision of an archival tumor sample to a Novartis designated laboratory for molecular profiling. The tumor material submitted for these analyses may have been obtained at any time during the course of the patient's disease.
4. Measurable disease as assessed by RECIST 1.1 for non-GBM tumors and by RANO criteria for GBM.
5. ECOG (WHO) performance status 0-2
6. Adequate bone marrow and organ function
7. Patient is able to swallow and retain oral medication
8. Negative serum pregnancy test; non-lactating or post-menopausal women.

Exclusion Criteria:

1.Use of other investigational drugs within 30 days of enrollment or 5 half-lives of enrollment, whichever is longer. 2.History of hypersensitivity to LDE225, BKM120 or to drugs of similar chemical classes.

3.Patient has received previous treatment with PI3K inhibitors and/or smoothened inhibitors.

4.Patients with recurrent GBM who have received radiotherapy within 3 months of initiating study treatment.

5.Patients with primary CNS tumor (except recurrent GBM), uncontrolled or symptomatic CNS metastasis. However, patients with controlled, asymptomatic or with resected CNS metastases with no radiological evidence of disease or with stable brain metastasis with no progression may be are eligible.

6.Patients who have neuromuscular disorders or are on concomitant treatment with drugs that are recognized to cause rhabdomyolysis, such as HMG CoA inhibitors (statins), clofibrate and gemfibrozil. If it is essential that the patient remains on a statin to control hyperlipidemia, only Pravastatin may be used with extra caution.

7.Patients who require the use of warfarin (substrate of CYP2C9) cannot be enrolled as LDE225 and BKM120 are competitive inhibitors of CYP2C9 based on in-vitro data.

8.Patient is currently being treated with drugs known to be strong inhibitors or inducers of CYP3A4/5, which cannot be discontinued or switched to a different medication 7 days prior to starting study treatment and for the duration of the study.

9.Patient has a score ≥12 on the PHQ-9 questionnaire. A normal evaluation by a psychiatrist or psychologist can overrule this exclusion).

10.Patients who select responses of "1", "2" or "3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9), (a normal evaluation by a psychiatrist or psychologist can overrule this exclusion).

11.Patient has a GAD-7 mood scale score ≥ 15, (a normal evaluation by a psychiatrist or psychologist can overrule this exclusion) 12.Patient has a documented medical history of or active major depression episode, bipolar disorder (I or II), obsessive compulsive disorder, schizophrenia, a history of suicidal attempts or ideation, or homicidal ideation (e.g. risk of doing harm to self or others) 13. Patient has ≥CTCAE grade 3 anxiety 14.Current medical history of the following:

* Use of a pacemaker
* History of or presence of clinically significant ventricular or atrial tachyarrhythmia
* Clinically significant resting bradycardia (< 45 beats per minute)
* History of clinically documented myocardial infarction
* History of unstable angina pectoris
* History of known structural abnormalities (i.e. cardiomyopathy) 15.Clinically significant cardio-vascular disease 16.Clinically significant abnormal ECG 17.Left Ventricular Ejection Fraction (LVEF) <50% as determined by Multiple Gated Acquisition (MUGA) scan or echocardiogram (ECHO) 18.Patient is currently receiving treatment with QT prolonging medication known to have a risk to induce Torsades de Pointes, and the treatment cannot be discontinued or switched to a different medication 7 days prior to starting the study and for the duration of the study 19.Patients who are not willing to apply highly effective contraception as defined by the protocol during the study and through the duration of the study. Note: Hormonal contraception methods (e.g. oral, injected, implanted) are not allowed as it cannot be ruled out that the study drug decreases the effectiveness of hormonal contraception 20.Sexually active males who are unwilling to use a condom during intercourse while taking drug and for 6 months after stopping investigational medications and agree not father a child in this period.

  21.Patients is currently receiving increasing or chronic treatment with corticosteroids ((≥ the anti-inflammatory potency of 4mg dexamethasone) or another immunosuppressive agent.

  22.Patient has been treated with any hematopoietic colony-stimulating growth factors (e.g., G-CSF, GM-CSF) ≤ 2 weeks prior to starting study drug. Erythropoietin or darbepoetin therapy, if initiated before enrollment, may be continued 23.Patient who has received chemotherapy, targeted therapy or immunotherapy ≤ 3 weeks (6 weeks for nitrosourea, mitomycin-C or monoclonal antibodies; 1 week for hormonal anti-cancer therapy) prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia, bone marrow and organ functions) 24.Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of LDE225 and BKM120 (e.g., ulcerative colitis, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection) 25.Patient has a known history of HIV infection (testing not mandatory)

AMENDMENT 1 CHANGES:

Inclusion Criteria:

3. Provision of an archival tumor sample to a Novartis designated laboratory for molecular profiling. It is accepted that it may not be possible to obtain all samples prior to commencing study treatment. It is also accepted that it may not be possible to obtain a sample (e.g. if sufficient sample does not exist), and in this situation inclusion of the patient should be discussed with Novartis (as this may not make a patient ineligible).

Exclusion Criteria:

5. Patients with primary CNS tumor (except recurrent GBM), uncontrolled or symptomatic CNS metastasis. However, patients with controlled, asymptomatic or with resected CNS metastases with no radiological evidence of disease or with stable brain metastasis with no progression may be eligible. The patient must have completed any prior treatment for CNS metastases (including radiotherapy and/or surgery) ≥ 28 days (> 14 days for stereotactic radiosurgery).

9. Patient has a score ≥12 on the PHQ-9 questionnaire. A normal evaluation by a psychiatrist can overrule this exclusion.

10.Patients who select responses of "1", "2" or "3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9), (a normal evaluation by a psychiatrist can overrule this exclusion).

11.Patient has a GAD-7 mood scale score ≥ 15, (a normal evaluation by a psychiatrist can overrule this exclusion)

AMENDMENT 2 CHANGES:

Updated Inclusion Criteria:

3. Revised to specify the groups of patients that will be included in the dose escalation and dose expansion parts (NEW tumor type added here): Patients with histologically/cytologically confirmed diagnosis of the following advanced tumors that have progressed despite standard therapy or that have no available established treatments: four group of patients during the dose escalation part: metastatic breast cancer, advanced pancreatic adenocarcinoma, metastatic CRC or recurrent GBM and five groups during the dose expansion part: triple negative metastatic breast cancer, hormone receptor positive (ER+/PR+, and Her2-) metastatic breast cancer, recurrent GBM, GASTRIC/GASTROESOPHAGEAL JUNCTION CANCER, advanced pancreatic adenocarcinoma or metastatic CRC will be included.

6. ECOG (WHO) performance status 0-2. ADDED "only applies to patients enrolled under the original and Amendment 1 protocol versions." 7. Two sub-bullets updated: Potassium, and calcium, within normal limits for the institution. Out of range values should be clinically insignificant. Serum Creatinine ≤ 1.5 x ULN and 24-hour creatinine clearance ≥ 50 mL/min (determined by inputting the serum creatinine result into the Cockcroft-Gault formula).

9. NEW Inclusion criterion: Recurrent GBM patient has a Karnofsky performance status (KPS) score ≥ 70.

10. NEW Inclusion criterion:ECOG (WHO) performance status 0-1 (only applies to patients enrolled under Amendment 2 and any later protocol versions).

Updated Exclusion Criteria:

12. Patient has a score ≥12 on the PHQ-9 questionnaire. REMOVED "A normal evaluation by a psychiatrist can overrule this exclusion." 13.Patients who select responses of "1", "2" or "3" to question number 9 on the PHQ-9 questionnaire regarding potential for suicidal thoughts or ideation (independent of the total score of the PHQ-9). REMOVED "A normal evaluation by a psychiatrist can overrule this exclusion." 14. Patient has a GAD-7 mood scale score ≥ 15. REMOVED "A normal evaluation by a psychiatrist can overrule this exclusion." 15. Patient has a documented medical history of or active major depression episode, bipolar disorder (I or II), obsessive compulsive disorder, schizophrenia, a history of suicidal attempts or ideation. ADDED "or homicidal ideation (e.g. risk of doing harm to self or others), or patients with active severe personality disorders (defined according to DSM- IV, Diagnostic and Statistical Manual of Mental Disorders, 4th edition) are not eligible. Note: for patients with psychotropic treatments ongoing at baseline, the dose and the schedule should not be modified within the previous 6 weeks prior to start of study drug." 23. REMOVED mention of "Double barrier method" term under "Male patient" section 27. Patient who has received chemotherapy, targeted therapy or immunotherapy ≤ 3 weeks (6 weeks for nitrosourea, or mitomycin-C; or 6 weeks for monoclonal antibodies if carryover effects are suspected; 1 week for hormonal anti-cancer therapy) prior to starting study drug or who have not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia, bone marrow and organ functions). ADDED clarification concerning the washout period for monoclonal antibodies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2012-07; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities | 6 weeks (42 days)
  Dose Limiting Toxicities (DLTs) during the first 6 weeks (42 days) of the combination treatment of LDE225 and BKM120.

SECONDARY OUTCOMES:
Number of Patients with Adverse Events and Serious Adverse Events | Following signing of the informed consent form, up to and including 30 days following the last dose
  Adverse and serious adverse events, changes in hematology and chemistry values, and assessment of physical and/or neurological examinations, vital signs, and electrocardiograms
Objective response rate (ORR) | 4 months
  ORR is the proportion of patients with best overall response of complete or partial response. ORR will be used to evaluate preliminary efficacy of the combination therapy. Tumors will be assessed using Investigator read CT/MRI assessments evaluated as per RECIST 1.1, except for patients with glioblastoma multiforme (GBM) who will be assessed per the RANO Criteria.
Early progression rate (EPR) | 6 months
  EPR is the proportion of patients with progressive disease within 6 months of the start of treatment. EPR will be used to evaluate preliminary efficacy of the combination therapy. Tumors will be assessed using Investigator read CT/MRI assessments evaluated as per RECIST 1.1, except for patients with GBM who will be assessed per the RANO Criteria. AMENDMENT #2 change: EPR duration modified to 6 months for recurrent GBM patients per the convention for that tumor type
Plasma pharmacokinetics (PK) parameters | In 28-day cycles: Cycle 1/Day 1 and Day 15; Cycle 2/Day 1 and Day 15; then on Day 1 of each additional cycle up to and including cycle 11 (if applicable)
  Plasma PK parameters of LDE225 and plasma PK parameters of BKM120.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmceuticals
Locations (22):
- United States (13):
  - Cedars Sinai Medical Center SC, Los Angeles, California
  - University of California San Francisco UCSF (SC), San Francisco, California
  - H. Lee Moffitt Cancer Center & Research Institute Moffitt 4, Tampa, Florida
  - Dana Farber Cancer Institute Dana SC, Boston, Massachusetts
  - Mayo Clinic - Rochester Division of Hematology, Rochester, Minnesota
  - Duke University Medical Center Duke - Baker, Durham, North Carolina
  - Willamette Valley Clinical Studies Williamette Valley Cancer, Eugene, Oregon
  - Northwest Cancer Specialists Northwest Cancer, Portland, Oregon
  - Fox Chase Cancer Center FCCC, Philadelphia, Pennsylvania
  - Texas Oncology Midtown Texas Oncology, Dallas, Texas
  - Sammons Cancer Center - Texas Oncology SC-2, Dallas, Texas
  - University of Texas/MD Anderson Cancer Center SC-3, Houston, Texas
  - University of Utah / Huntsman Cancer Institute Huntsman, Salt Lake City, Utah
- Novartis Investigative Site, Parkville, Victoria, Australia
- Novartis Investigative Site, Wilrijk, Belgium
- Novartis Investigative Site, Edmonton, Alberta, Canada
- Novartis Investigative Site, Essen, Germany
- Italy (2):
  - Novartis Investigative Site, Ancona, AN
  - Novartis Investigative Site, Milan, MI
- Novartis Investigative Site, Barcelona, Catalonia, Spain
- United Kingdom (2):
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Sutton

REFERENCES:
- See also: Results for CLDE225X2114 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=14654